CLINICAL TRIAL: NCT05347485
Title: A Safety and Efficacy Study of JNJ-68284528 (Ciltacabtagene Autoleucel) Out-of-Specification (OOS) for Commercial Release in Patients With Multiple Myeloma
Brief Title: A Study of JNJ-68284528 Out-of-Specification (OOS) for Commercial Release in Participants With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR109014; 68284528MMY2005 (Other: Janssen Research & Development, LLC)
Expanded Access: NCT05346835 (Available)
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ciltacabtagene Autoleucel (Cilta-cel) (Experimental): Eligible participants will receive bridging therapy (that is, anti-plasma cell directed treatment) based on participant's clinical status and timing of availability of cilta-cel (JNJ-68284528) along with lymphodepleting chemotherapy (cyclophosphamide 300 milligrams per meter square [mg/m^2] intravenous [IV] and fludarabine 30 mg/m^2 IV daily, for 3 days). After 5 to 7 days of initiating lymphodepleting chemotherapy, participants will receive a single IV infusion of cilta-cel (JNJ-68284528) at a total targeted dose of 0.75*10^6 chimeric antigen receptor (CAR)-positive viable T cells per kilogram (cells/kg).
  Interventions: Drug: Cilta-cel; Drug: Lymphodepleting Therapy (Cyclophosphamide and Fludarabine)

INTERVENTIONS:
Drug: Cilta-cel — Cilta-cel will be administered as an IV infusion.
  Other Names: JNJ-68284528
Drug: Lymphodepleting Therapy (Cyclophosphamide and Fludarabine) — Lymphodepleting therapy (cyclophosphamide and fludarabine) will be administered intravenously.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of cilta-cel out-of-specification (OOS).

ELIGIBILITY:
Inclusion Criteria:

* Eligible for treatment with cilta-cel per United States prescribing information (USPI) or locally approved label
* Participant is suffering from serious or life threatening multiple myeloma per USPI (or locally approved label, respectively), and re-apheresis, re-manufacturing, or other anti-myeloma directed therapies is not considered feasible or adequate per investigator
* Has adequate general health status and organ function per investigator assessment and meets the criteria to receive cilta-cel out-of-specifications (OOS)
* Meets the criteria to receive lymphodepleting chemotherapy
* A woman of childbearing potential must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) pregnancy test during screening and prior to the first dose of cyclophosphamide and fludarabine

Exclusion Criteria:

* History of active uncontrolled infection or condition where an administration of cilta-cel OOS constitutes serious health risk to the participant
* Known allergies, hypersensitivity, or intolerance to the excipients of cilta-cel OOS including dimethyl sulfoxide (DMSO), dextran 40, or residual kanamycin per USPI
* Hepatitis B infection
* Hepatitis C infection defined as (anti hepatitis C virus [HCV] antibody positive or detectable HCV ribonucleic acid [RNA]) or known to have a history of hepatitis C
* Seropositive for human immunodeficiency virus (HIV)
* Uncontrolled autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (18):
- United States (18):
  - City of Hope, Duarte, California
  - University of California San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Kansas University Medical Center, Westwood, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Medical College Of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS): Adult participants aged 18 years or older, with multiple myeloma received the lymphodepleting chemotherapy (cyclophosphamide 300 milligrams per meter square [mg/m^2] intravenous [IV] infusion and fludarabine 30 mg/m^2 IV infusion daily, for 3 days [Day -7 to Day -5]). After 5 to 7 days of initiating lymphodepleting chemotherapy, participants received IV infusion of cilta-cel OOS at a total targeted dose of 0.75*10^6 chimeric antigen receptor (CAR)-positive viable T-cells/kg (dose range 0.5*10^6 CAR-positive viable T cells/kg to 1.0*10^6 CAR-positive viable T cells/kg) based on participant's body weight at apheresis or per exceptional release criteria determined alternative dose.
Period: Overall Study
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Started | 86
Treated | 82
Completed | 0
Not Completed | 86
Not completed — Death | 14
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 13
Not completed — Progressive Disease | 1
Not completed — Study Terminated by Sponsor | 49
Not completed — Other | 1
Not completed — Enrolled (consented) but not treated | 4
Not completed — Disease Relapse | 2

BASELINE CHARACTERISTICS:
Population: The all treated analysis set included all participants who received study intervention (cilta-cel out-of-specifications [OOS]).
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 76
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 55
  More than one race | 1
  Unknown or Not Reported | 10
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 82

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of participants who had partial response (PR) or better (sCR+CR+VGPR+PR) according to the International Myeloma Working Group (IMWG) response criteria, as assessed by the investigator. CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and less than (<) 5 percentage (%) plasma cells (PCs) in bone marrow; sCR: CR+Normal free light chain ratio and absence of clonal cells in bone marrow by immunohistochemistry or immuno fluorescence; PR: greater than equal to (>=) 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >= 90 percentage (%) or to <200 mg/24 hours; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 mg per 24 hour.
Time Frame: From Day 1 (post infusion) up to 18.6 months
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Percentage of participants | 57.3 [45.9 to 68.2]

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs were reported. An AE was any untoward medical occurrence in a participant participating in a clinical study that did not necessarily had a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as any AE that occurred on or after the start of cilta-cel OOS infusion through 100 days after the cilta-cel OOS infusion or the start of subsequent anti-myeloma therapy, whichever was earlier; or any AE that was considered related to study intervention regardless of the start date of the event; or any AE that was present at baseline (Day 1, infusion of cilta-cel OOS) but worsens in toxicity grade or is subsequently considered related to study intervention by the investigator.
Time Frame: From Day 1 up to 100 days post cilta-cel OOS infusion (Up to 100 days)
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS).
Measure: Count of Participants; unit: Participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Participants | 81

3. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) by Severity
Description: An AE was any untoward medical occurrence in a participant participating in a clinical study that did not necessarily had a causal relationship with the pharmaceutical/biological agent under study. TEAEs were defined as any AE that occurs on or after the start of cilta-cel OOS infusion through 100 days after the cilta-cel OOS infusion or the start of subsequent anti-myeloma therapy, whichever was earlier; or any AE that is considered related to study intervention regardless of the start date of the event; or any AE that was present at baseline (Day 1, pre-infusion of cilta-cel OOS) but worsens in toxicity grade or was subsequently considered related to study intervention by the investigator. Severity was assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 as: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death related to adverse event.
Time Frame: From Day 1 up to 100 days post cilta-cel OOS infusion (Up to 100 days)
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS).
Measure: Count of Participants; unit: Participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Participants
  Grade 1: Mild | 1
  Grade 2: Moderate | 6
  Grade 3: Severe | 14
  Grade 4: Life-threatening | 51
  Grade 5: Death | 9

4. Secondary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: Number of participants with serious TESAEs were reported. A SAE was defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly/birth defect in the offspring of a participant, or was an important medical event. TESAEs were defined as any SAE that occurs on or after the start of cilta-cel OOS infusion through 100 days after the cilta-cel OOS infusion or the start of subsequent anti-myeloma therapy, whichever was earlier; or any SAE that was considered related to study intervention regardless of the start date of the event; or any SAE that was present at baseline but worsens in toxicity grade or was subsequently considered related to study intervention by the investigator.
Time Frame: From Day 1 up to 100 days post cilta-cel OOS infusion (Up to 100 days)
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS).
Measure: Count of Participants; unit: Participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Participants | 42

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Event of Special Interest (AESIs): Cytokine Release Syndrome (CRS), Immune Effector Cell-Associated Neurotoxicity (ICANS), Other Neurotoxicities, and Secondary Primary Malignancies
Description: Number of participants with treatment-emergent AESIs: CRS, ICANS, other neurotoxicities, and secondary primary malignancies were reported. AESIs include the anticipated risks of treatment with study drug and events that may be related to multiple sclerosis comorbidities. Treatment-emergent AESIs were defined as any AESI that occurs on or after the start of cilta-cel OOS infusion through 100 days after the cilta-cel OOS infusion or the start of subsequent anti-myeloma therapy, whichever was earlier; or any AESI that was considered related to study intervention regardless of the start date of the event; or any AESI that was present at baseline but worsens in toxicity grade or was subsequently considered related to study intervention by the investigator.
Time Frame: From Day 1 up to 100 days post cilta-cel OOS infusion (Up to 100 days)
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS).
Measure: Count of Participants; unit: Participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Participants
  Cytokine Release Syndrome (CRS) | 61
  Immune Effector Cell-Associated Neurotoxicity (ICANS) | 12
  Other neurotoxicities | 8
  Secondary primary malignancies | 5

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Event of Special Interest (AESIs): Prolonged and Recurrent Cytopenias
Description: Number of participants with treatment-emergent AESIs: prolonged and recurrent cytopenias were reported. AESIs include the anticipated risks of treatment with study drug and events that may be related to multiple sclerosis comorbidities. It included Thrombocytopenia, Neutropenia, Lymphopenia, and Anaemia. Treatment-emergent AESIs were defined as any AESI that occurs on or after the start of cilta-cel OOS infusion through 100 days after the cilta-cel OOS infusion or the start of subsequent anti-myeloma therapy, whichever was earlier; or any AESI that was considered related to study intervention regardless of the start date of the event; or any AESI that was present at baseline but worsens in toxicity grade or was subsequently considered related to study intervention by the investigator. Severity was assessed using NCI-CTCAE version 5.0 as: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; Grade 5: Death related to adverse event.
Time Frame: From Day 1 up to 100 days post cilta-cel OOS infusion (Up to 100 days)
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS).
Measure: Count of Participants; unit: Participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Participants
  Thrombocytopenia: Grade 3/4 After Day 1 Dosing | 50
  Thrombocytopenia: Initial Grade 3/4 Not Recovered to <= Grade 2 by Day 30 | 42
  Thrombocytopenia: Initial Grade 3/4 Not Recovered to <= Grade 2 by Day 60 | 29
  Thrombocytopenia: Grade 3/4 > Day 60 (After Initial Recovery of Grade 3/4 within Day 60) | 1
  Neutropenia: Grade 3/4 After Day 1 Dosing | 75
  Neutropenia: Initial Grade 3/4 Not Recovered to <= Grade 2 by Day 30 | 36
  Neutropenia: Initial Grade 3/4 Not Recovered to <= Grade 2 by Day 60 | 18
  Neutropenia: Grade 3/4 > Day 60 (After Initial Recovery of Grade 3/4 within Day 60) | 1
  Lymphopenia: Grade 3/4 After Day 1 Dosing | 75
  Lymphopenia: Initial Grade 3/4 Not Recovered to <= Grade 2 by Day 30 | 32
  Lymphopenia: Initial Grade 3/4 Not Recovered to <= Grade 2 by Day 60 | 21
  Lymphopenia: Grade 3/4 > Day 60 (After Initial Recovery of Grade 3/4 within Day 60) | 4
  Anaemia: Grade 3/4 After Day 1 Dosing | 36
  Anaemia: Initial Grade 3/4 Not Recovered to <= Grade 2 by Day 30 | 12
  Anaemia: Initial Grade 3/4 Not Recovered to <= Grade 2 by Day 60 | 9
  Anaemia: Grade 3/4 > Day 60 (After Initial Recovery of Grade 3/4 within Day 60) | 2

7. Secondary Outcome: Number of Participants by Worst Grade Abnormalities in Clinical Laboratory Tests: Hematology (Including Coagulation) and Chemistry After Cilta-cel OOS Infusion
Description: Number of participants by worst grade abnormalities in clinical laboratory tests: hematology (including coagulation) and chemistry, after cilta-cel OOS infusion were reported. Grades were assessed using NCI-CTCAE (version 5.0), as: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening. Participants with normal values or a value in the opposite direction (for laboratory tests with bidirectional toxicities defined) were assigned Grade 0. Only those categories in which at least 1 participant had data were reported.
Time Frame: From Day 1 (post infusion) up to 18.6 months
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS). Here, 'N' (number of participants analyzed) signifies number of participants analyzed for this outcome measure. Here, 'n' (number analyzed) signifies number of participants analyzed for each specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 81
Participants
  Hematology: Activated partial thromboplastin time prolonged: Grade 0: number analyzed (Participants) | 2
  Hematology: Activated partial thromboplastin time prolonged: Grade 0 | 1
  Hematology: Activated partial thromboplastin time prolonged: Grade 2: number analyzed (Participants) | 2
  Hematology: Activated partial thromboplastin time prolonged: Grade 2 | 1
  Hematology: Hemoglobin (Anemia): Grade 1 | 9
  Hematology: Hemoglobin (Anemia): Grade 2 | 33
  Hematology: Hemoglobin (Anemia): Grade 3 | 39
  Hematology: Lymphocyte count decreased: Grade 0 | 3
  Hematology: Lymphocyte count decreased: Grade 1 | 1
  Hematology: Lymphocyte count decreased: Grade 2 | 2
  Hematology: Lymphocyte count decreased: Grade 3 | 10
  Hematology: Lymphocyte count decreased: Grade 4 | 65
  Hematology: Neutrophil count decreased: Grade 0 | 1
  Hematology: Neutrophil count decreased: Grade 1 | 1
  Hematology: Neutrophil count decreased: Grade 2 | 4
  Hematology: Neutrophil count decreased: Grade 3 | 21
  Hematology: Neutrophil count decreased: Grade 4 | 54
  Hematology: Platelet count decreased: Grade 0 | 1
  Hematology: Platelet count decreased: Grade 1 | 16
  Hematology: Platelet count decreased: Grade 2 | 14
  Hematology: Platelet count decreased: Grade 3 | 15
  Hematology: Platelet count decreased: Grade 4 | 35
  Hematology: White blood cell decreased: Grade 2 | 4
  Hematology: White blood cell decreased: Grade 3 | 21
  Hematology: White blood cell decreased: Grade 4 | 56
  Biochemistry: Alanine Aminotransferase increased: Grade 0 | 53
  Biochemistry: Alanine Aminotransferase increased: Grade 1 | 20
  Biochemistry: Alanine Aminotransferase increased: Grade 2 | 5
  Biochemistry: Alanine Aminotransferase increased: Grade 3 | 3
  Biochemistry: Aspartate aminotransferase increased: Grade 0 | 43
  Biochemistry: Aspartate aminotransferase increased: Grade 1 | 28
  Biochemistry: Aspartate aminotransferase increased: Grade 2 | 5
  Biochemistry: Aspartate aminotransferase increased: Grade 3 | 4
  Biochemistry: Aspartate aminotransferase increased: Grade 4 | 1
  Biochemistry: Alkaline phosphatase high: Grade 0 | 58
  Biochemistry: Alkaline phosphatase high: Grade 1 | 18
  Biochemistry: Alkaline phosphatase high: Grade 2 | 4
  Biochemistry: Alkaline phosphatase high: Grade 3 | 1
  Biochemistry: Blood bilirubin increased: Grade 0 | 63
  Biochemistry: Blood bilirubin increased: Grade 1 | 6
  Biochemistry: Blood bilirubin increased: Grade 2 | 9
  Biochemistry: Blood bilirubin increased: Grade 3 | 2
  Biochemistry: Blood bilirubin increased: Grade 4 | 1
  Biochemistry: Hypercalcemia: Grade 0 | 76
  Biochemistry: Hypercalcemia: Grade 1 | 4
  Biochemistry: Hypercalcemia: Grade 2 | 1
  Biochemistry: Hypocalcemia: Grade 0 | 36
  Biochemistry: Hypocalcemia: Grade 1 | 23
  Biochemistry: Hypocalcemia: Grade 2 | 19
  Biochemistry: Hypocalcemia: Grade 4 | 3
  Biochemistry: Creatinine increased: Grade 0 | 53
  Biochemistry: Creatinine increased: Grade 1 | 16
  Biochemistry: Creatinine increased: Grade 2 | 7
  Biochemistry: Creatinine increased: Grade 3 | 3
  Biochemistry: Creatinine increased: Grade 4 | 2

8. Secondary Outcome: Partial Response (PR) Rate
Description: PR rate was defined as percentage of participants who achieved PR according to IMWG response criteria. PR was defined as per IMWG criteria as >= 50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >= 90% or to < 200 mg/24hours. If the serum and urine M-protein were unmeasurable, a >= 50% decrease in the difference between involved and uninvolved Free light chain (FLC) levels was required in the place of the M-protein criteria. If serum and urine M-protein were not measurable, and serum free light assay was also not measurable, >=50% reduction in bone marrow plasma cells is required in place of M-protein, provided baseline bone marrow plasma cells percentage was >=30%. In addition to the above listed criteria, if present at baseline, a >= 50% reduction in the size of soft tissue plasmacytomas was also required.
Time Frame: From Day 1 (post infusion) up to 18.6 months
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Percentage of Participants | 9.8 [4.3 to 18.3]

9. Secondary Outcome: Very Good Partial Response (VGPR) Rate
Description: VGPR rate is defined as percentage of participants who achieved best response of VGPR according to IMWG response criteria. As per IMWG response criteria, VPGR: serum and urine M-component detectable by immunofixation but not on electrophoresis, or >=90% reduction in serum M-component plus urine M-component <100 mg/24 hours.
Time Frame: From Day 1 (post infusion) up to 18.6 months
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Percentage of Participants | 14.6 [7.8 to 24.2]

10. Secondary Outcome: Complete Response (CR) Rate
Description: CR rate is defined as percentage of participants who achieved best response of CR according to IMWG response criteria. CR is defined as per IMWG criteria as negative immunofixation of serum and urine, and disappearance of any soft tissue plasmacytomas, and <5% PCs in bone marrow. No evidence of initial monoclonal protein isotype(s) on immunofixation of the serum and urine.
Time Frame: From Day 1 (post infusion) up to 18.6 months
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Percentage of Participants | 17.1 [9.7 to 27.0]

11. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical benefit rate was defined as the percentage of participants who achieved a minimal response (MR) or better (including MR, PR, VGPR, CR, and sCR). MR was defined as per IMWG criteria as >=25% but less than or equal to (<=) 49% reduction of serum M-protein and reduction in 24-hour urine M-protein by 50% to 89%. In addition to the above criteria, if present at baseline, >=50% reduction in the size of soft tissue plasmacytomas was also required.
Time Frame: From Day 1 (post infusion) up to 18.6 months
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Percentage of Participants | 59.8 [48.3 to 70.4]

12. Secondary Outcome: Stringent Complete Response (sCR) Rate
Description: sCR rate is defined as percentage of participants who achieved sCR according to IMWG response criteria. sCR is defined per IMWG criteria as CR plus normal FLC ratio, and absence of clonal PCs by immunohistochemistry or 2- to 4-color flow cytometry. CR is defined as per IMWG as negative immunofixation of serum and urine, and disappearance of any soft tissue plasmacytomas, and <5% PCs in bone marrow. No evidence of initial monoclonal protein isotype(s) on immunofixation of the serum and urine.
Time Frame: From Day 1 (post infusion) up to 18.6 months
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Percentage of Participants | 15.9 [8.7 to 25.6]

13. Secondary Outcome: Duration of Response (DOR)
Description: DOR calculated in responders (with PR or better response) from date of initial documentation of response (PR or better) to date of first documented evidence of progressive disease (PD) as per IMWG criteria, or death due to any cause, whichever occurs first. PD: increase of 25% from lowest response value: serum and urine M-component (absolute increase must be >=0.5 grams/deciliter [g/dL] and >=200 mg/24 hours, respectively); only in participants without measurable serum and urine M-protein levels, difference between involved and uninvolved FLC levels (absolute increase must be >10 mg/dL); only in participants without measurable serum and/or urine M-protein levels and without measurable disease by FLC levels, bone marrow PC % (absolute increase must be >=10%), appearance of new lesion; definite development of new bone lesions or definite increase in the size of existing bone lesions, >=50% increase in circulating PCs (minimum of 200 cells per uL) if this was the only measure of disease.
Time Frame: From Day 1 (post infusion) up to 18.6 months
Population: Analysis population included responders (who achieved PR or better response) in all treated analysis set. The all treated analysis set included all participants who received study intervention (cilta-cel OOS). Here, 'N' (number of participants analyzed) signifies number of participants analyzed for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 47
Months | NA [7.75 to NA] — Median and upper limit of 95% CI could not be estimated due to low number of participants with events.

14. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS defined as the time from the date of the initial infusion of cilta-cel OOS to the date of first documented disease progression as per IMWG criteria, or death due to any cause, whichever occurs first. PD: increase of 25% from lowest response value: serum and urine M-component (absolute increase must be >=0.5 g/dL and >=200 mg/24 hours, respectively); only in participants without measurable serum and/or urine M-protein levels the difference between involved and uninvolved FLC levels (absolute increase must be >10 mg/dL); only in participants without measurable serum and urine M-protein levels and without measurable disease by FLC levels, bone marrow PC percentage (absolute increase must be >=10%), appearance of a new lesion; definite development of new bone lesions or definite increase in the size of existing bone lesions, >=50% increase in circulating PCs (minimum of 200 cells per uL) if this was the only measure of disease.
Time Frame: From Day 1 (post infusion) up to 18.6 months
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Months | NA [7.39 to NA] — Median and upper limit of 95% CI could not be estimated due to low number of participants with events.

15. Secondary Outcome: Overall Survival (OS)
Description: OS is measured from the date of the initial infusion of cilta-cel OOS to the date of the participant's death. If the participant is alive or the vital status is unknown, then the participant's data was censored at the date the participant was last known to be alive.
Time Frame: From Day 1 (post infusion) up to 18.6 months
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 82
Months | NA [13.67 to NA] — Median and upper limit of 95% CI could not be estimated due to low number of participants with events.

16. Secondary Outcome: Minimal Residual Disease (MRD)-Negative Rate
Description: MRD-negative rate is defined as the percentage of participants with negative MRD status (at 10^-4, 10^-5 and 10^-6 cutoffs) by bone marrow aspirate.
Time Frame: From Day 1 (post infusion) up to 18.6 months
Population: All participants who received cilta-cel OOS and had evaluable MRD samples in all treated analysis set. The all treated analysis set included all participants who received study intervention (cilta-cel OOS). Here, 'N' (number of participants analyzed) signifies number of participants analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 15
Percentage of participants
  10^-4 cutoff | 66.7 [38.4 to 88.2]
  10^-5 cutoff | 66.7 [38.4 to 88.2]
  10^-6 cutoff | 53.3 [26.6 to 78.7]

17. Secondary Outcome: Number of Participants With Presence of Replication Competent Lentivirus
Description: Number of participants with presence of replication competent lentivirus (with evaluable sample) were reported.
Time Frame: Predose, 3, 6, 12 months after cilta-cel infusion on Day 1
Population: The all treated analysis set included all participants who received study intervention (cilta-cel OOS). Here, 'N' (number of participants analyzed) signifies number of participants analyzed for this outcome measure. Here, 'n' (number analyzed) signifies number of participants analyzed at each specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
Number analyzed (Participants) | 57
Participants
  Predose of cilta-cel infusion | 0
  3 months after cilta-cel infusion: number analyzed (Participants) | 26
  3 months after cilta-cel infusion | 0
  6 months after cilta-cel infusion: number analyzed (Participants) | 30
  6 months after cilta-cel infusion | 0
  12 months after cilta-cel infusion: number analyzed (Participants) | 12
  12 months after cilta-cel infusion | 0

ADVERSE EVENTS:
Time Frame: All-cause Mortality: From Day 1 (post infusion) up to 18.6 months; Serious and Other AEs: From Day 1 (post infusion) up to Day 100
Description: All-treated analysis set which included all participants who received study intervention (cilta-cel out-of-specifications [OOS]).
Arm/Group | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS)
All-Cause Mortality (participants affected / at risk) | 16/82
Serious Adverse Events (participants affected / at risk) | 42/82
Other Adverse Events (participants affected / at risk) | 81/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS) (N=82)
Anaemia (Blood and lymphatic system disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Adrenal Insufficiency (Endocrine disorders) | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 2
Pyrexia (General disorders) | 2
Cytokine Release Syndrome (Immune system disorders) | 19
Adenovirus Infection (Infections and infestations) | 1
Clostridium Difficile Colitis (Infections and infestations) | 1
Covid-19 (Infections and infestations) | 2
Cytomegalovirus Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 5
Septic Embolus (Infections and infestations) | 1
Septic Shock (Infections and infestations) | 1
Streptococcal Bacteraemia (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 3
Urinary Tract Infection (Infections and infestations) | 1
Liver Function Test Increased (Investigations) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Bell's Palsy (Nervous system disorders) | 3
Cerebral Haemorrhage (Nervous system disorders) | 1
Haemorrhage Intracranial (Nervous system disorders) | 2
Immune Effector Cell-Associated Neurotoxicity Syndrome (Nervous system disorders) | 8
Neurotoxicity (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Renal Tubular Necrosis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Haematoma (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ciltacabtagene Autoleucel (Cilta-cel) Out-of-Specification (OOS) (N=82)
Anaemia (Blood and lymphatic system disorders) | 49
Febrile Neutropenia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 44
Lymphopenia (Blood and lymphatic system disorders) | 26
Neutropenia (Blood and lymphatic system disorders) | 66
Thrombocytopenia (Blood and lymphatic system disorders) | 46
Atrial Fibrillation (Cardiac disorders) | 5
Sinus Bradycardia (Cardiac disorders) | 5
Sinus Tachycardia (Cardiac disorders) | 10
Dry Eye (Eye disorders) | 5
Vision Blurred (Eye disorders) | 5
Abdominal Pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 25
Nausea (Gastrointestinal disorders) | 26
Stomatitis (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 27
Oedema Peripheral (General disorders) | 10
Pain (General disorders) | 5
Pyrexia (General disorders) | 10
Hyperbilirubinaemia (Hepatobiliary disorders) | 7
Cytokine Release Syndrome (Immune system disorders) | 47
Hypogammaglobulinaemia (Immune system disorders) | 11
Covid-19 (Infections and infestations) | 7
Upper Respiratory Tract Infection (Infections and infestations) | 6
Urinary Tract Infection (Infections and infestations) | 5
Activated Partial Thromboplastin Time Prolonged (Investigations) | 5
Alanine Aminotransferase Increased (Investigations) | 11
Aspartate Aminotransferase Increased (Investigations) | 19
Blood Alkaline Phosphatase Increased (Investigations) | 8
Blood Creatinine Increased (Investigations) | 10
Blood Fibrinogen Decreased (Investigations) | 7
Blood Lactate Dehydrogenase Increased (Investigations) | 9
Gamma-Glutamyltransferase Increased (Investigations) | 9
Decreased Appetite (Metabolism and nutrition disorders) | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 6
Hyperphosphataemia (Metabolism and nutrition disorders) | 6
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 11
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 18
Hypokalaemia (Metabolism and nutrition disorders) | 19
Hypomagnesaemia (Metabolism and nutrition disorders) | 15
Hyponatraemia (Metabolism and nutrition disorders) | 17
Hypophosphataemia (Metabolism and nutrition disorders) | 24
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back Pain (Musculoskeletal and connective tissue disorders) | 7
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 19
Immune Effector Cell-Associated Neurotoxicity Syndrome (Nervous system disorders) | 9
Paraesthesia (Nervous system disorders) | 5
Tremor (Nervous system disorders) | 6
Confusional State (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 14
Acute Kidney Injury (Renal and urinary disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 11
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 5
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5
Flushing (Vascular disorders) | 5
Hypertension (Vascular disorders) | 11
Hypotension (Vascular disorders) | 13
Orthostatic Hypotension (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/85/NCT05347485/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT05347485/SAP_001.pdf